CLINICAL TRIAL: NCT05810558
Title: Impact of Glycine-augmented Prophylaxis on Resolution of Peri-implant Mucositis
Brief Title: Impact of Glycine Therapy on Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016H0397
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Ultrasonic (Placebo Comparator): Subjects will receive cleaning of the peri-implant sulcus using ultrasonic instrumentation
  Interventions: Procedure: Ultrasonic instrumentation
- Arm 2 Glycine (Experimental): Subjects will receive cleaning of the peri-implant sulcus using glycine powder air-powered debridement
  Interventions: Procedure: glycine powder air-powered debridement

INTERVENTIONS:
Procedure: glycine powder air-powered debridement — The intervention treatment consist sof glycine powder air-abrasive debridement (GPAD) using a handheld air polishing device, disposable subgingival nozzle, and glycine powder The nozzle is inserted to the depth of the pocket and all surfaces of the implant (mesial, buccal, distal, lingual) debrided for 5 seconds.
  Arms: Arm 2 Glycine
Procedure: Ultrasonic instrumentation — The control treatment consists of supragingival and root debridement using an ultrasonic scaler on low-medium power and coronal polishing with fine grit paste
  Arms: Arm 1 Ultrasonic

SUMMARY:
The purpose of this research study is to determine the impact of glycine powder air-abrasive debridement (GPAD) on the microbiology of the tissues surrounding dental implants with health and inflammation (peri-implant mucositis).

DETAILED DESCRIPTION:
Peri-implant mucositis, or the infection of the gingival tissues surrounding a dental implant, and peri-implantitis, or the infection of the gingival tissue surrounding a dental implant with bone loss, can lead to the failure and eventual loss of dental implants. The prevalence of peri-implant mucositis ranges from 30.7-43% and the prevalence of peri-implantitis ranges from 9.6-22% with non-smokers. Traditional treatment of this disease has been through biofilm removal using ultrasonic instrumentation. Glycine is a non-essential amino acid that possesses an anti-inflammatory, immunomodulary, and a cytoprotective effect. The goal of this investigation is to examine the impact of glycine-augmented biofilm removal on resolution of peri-implant mucositis

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Must have >1 tooth-borne, non-splinted single dental implant
* Signs of healthy dental implants (pocket probing depth <4mm and a lack of bleeding upon probing at peri-implant site) OR
* Signs of peri-implant mucositis (> 4mm probing pocket depths at the dental implant site, bleeding upon probing at >1 peri-implant site, pre-brushing plaque score of > 1.9 (modified Plaque Index (mPI)), and radiographic evidence of bone loss less than 2mm).

Exclusion Criteria:

* Uncontrolled medical condition (i.e. Diabetes, History of smoking <5 years)
* Pregnant or lactating females
* Untreated periodontal conditions
* Use of antibiotics in the past 3 months
* Subjects treated with medication for >2 weeks with known effects to the oral tissues (i.e. coumadin, phenytoin, nifedipine, cyclosporine, non-steroidal anti-inflammatory drugs)
* Signs of peri-implantitis (pocket probing depth of 4-6mm with bleeding upon probing at >1 peri-implant site AND radiographic bone loss)
* Dental implant mobility

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
gingival inflammation | 6 months
  presence of redness, bleeding on gentle probing from the peri-implant sulcus

CONTACTS AND LOCATIONS:
Overall Officials: Purnima S Kumar, DDS, PhD, Principal Investigator — Ohio State University
Locations (1):
- College of Dentistry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Partido B, Saraswat S, Kumar PS. Impact of Glycine Powder Air-Abrasive Debridement on Peri-Implant Mucositis: A Randomized Control Trial of Clinical, Microbial, and Immunological Changes. Clin Oral Implants Res. 2025 Jan;36(1):82-91. doi: 10.1111/clr.14361. Epub 2024 Sep 28. PMID 39340233